CLINICAL TRIAL: NCT03913091
Title: Liposomal Bupivacaine (Exparel ® ) Plus 0.5% Bupivacaine HCL Versus 0.5% Bupivacaine HCL for Interscalene Nerve Block (ISB) for Patients Undergoing Total Shoulder Arthroplasty(TSA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-01183
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Shoulder Pain
Keywords: Total Shoulder Arthroplasty (TSA); Interscalene Nerve Block (ISB)
MeSH Terms: conditions — Shoulder Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 20 mL 0.5% Bupivacaine HCL (Experimental)
  Interventions: Drug: 0.5% Bupivacaine HCL
- Interscalene nerve block with Liposomal + Bupivacaine 0.5% (Experimental): Administered in an Interscalene block for TSA
  Interventions: Drug: Liposomal Bupivacaine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Liposomal Bupivacaine Plus 0.5% Bupivacaine HCL
  Other Names: Exparel
  Arms: Interscalene nerve block with Liposomal + Bupivacaine 0.5%
Drug: 0.5% Bupivacaine HCL — 0.5% Bupivacaine HCL for Interscalene Nerve Block (ISB)
  Arms: 20 mL 0.5% Bupivacaine HCL

SUMMARY:
This is a phase IV , randomized, single-blind, single-center study comparing patient related outcomes such as postoperative pain and opioid usage for patients who receive ISB 's containing liposomal bupivacaine (Exparel®) plus 0.5% bupivacaine HCL versus 0.5% bupivacaine HCL undergoing total shoulder arthroplasty. The objective of this study is to compare opioid utilization and pain management of patients who receive Exparel in an ISB vs standard 0.5% bupivacaine HCL during the initial 72 --- hour post --- operative period. Additionally, to understand the duration of block after addition of Exparel® to bupivacaine in an Interscalene block after TSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total shoulder arthroplasty;
* Patients who consent to be randomized.

Exclusion Criteria:

* Patients younger than 18 and older than 75;
* Patients with a history of chronic pain that have used opioids for pain management for 3 months or longer;
* Patients who are allergic to oxycodone;
* Patients who are unable to speak English;
* Patients with diagnosed or self---reported cognitive dysfunction;
* Patients with a history of neurologic disorder that can interfere with pain sensation;
* Patients with a history of drug or recorded alcohol abuse;
* Patients who are unable to understand or follow instructions;
* Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease;
* Patients with an allergy or contraindication to any of the medications used in the study, or patients with a contraindication to any study procedures;
* Patients with BMI over 40;
* Any patient that the investigators feel cannot comply with all study related procedures;
* NYU Langone Health students, residents, faculty or staff members

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uchenna Umeh, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). Data will be available to achieve aims in the approved proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date
Access Criteria: Requests should be directed to uchenna.umeh@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.
  Access will be given to researchers who provide a methodologically sound proposal and investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 mL 0.5% Bupivacaine HCL | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5%
Started | 92 | 92
Completed | 72 | 78
Not Completed | 20 | 14
Not completed — Lost to Follow-up | 18 | 11
Not completed — Required additional meds/surgery | 1 | 2
Not completed — Chronic pain/history of substance abuse | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 mL 0.5% Bupivacaine HCL | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5% | Total
Number analyzed (Participants) | 72 | 78 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.39 (8.77) | 68.87 (8.83) | 67.63 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 39 | 69
  Male | 42 | 39 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 65 | 69 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 60 | 61 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 72 | 78 | 150

OUTCOME MEASURES:

1. Primary Outcome: Opioid Utilization
Description: Measure in morphine milligram equivalents [MME]
Time Frame: 24-72 hour, Post-Operative Period
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | 20 mL 0.5% Bupivacaine HCL | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5%
Number analyzed (Participants) | 72 | 78
Morphine Milligram Equivalents (MME) | 54.79 (15.26) | 30.38 (11.62)

2. Secondary Outcome: Opioid Utilization
Description: Measure in morphine milligram equivalents [MME]
Time Frame: Day 4-7, Post-Operative Period
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Arm/Group | 20 mL 0.5% Bupivacaine HCL | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5%
Number analyzed (Participants) | 72 | 78
Morphine Milligram Equivalents (MME) | 36.44 (11.13) | 18.73 (7.55)

3. Secondary Outcome: Score on Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Scale
Description: PROMIS Pain Intensity surveys are made up of three pain intensity questions, on a scale of 1-5.
  1. = No pain
  2. = Mild
  3. = Moderate
  4. = Severe
  5. = Very Severe
Time Frame: Day 1-7, Post-Operative Period
Population: The sample size is slightly smaller because this data was not collected at the beginning of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20 mL 0.5% Bupivacaine HCL | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5%
Number analyzed (Participants) | 67 | 72
score on a scale
  "In the past 7 days, how intense was your pain at its worst?" | 3.7 (1.16) | 3.07 (1.02)
  "In the past 7 days, how intense was your average pain?" | 2.81 (1.2) | 2.39 (1)
  "What is your level of pain right now?" | 2.22 (1.16) | 1.83 (1.02)

4. Secondary Outcome: T-Scores, PROMIS Pain Intensity Scale
Description: PROMIS Pain Intensity surveys are made up of three pain questions, which generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population.
Time Frame: Day 1-7, Post-Operative Period
Population: The sample size is slightly smaller because this data was not collected at the beginning of the study.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | 20 mL 0.5% Bupivacaine HCL | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5%
Number analyzed (Participants) | 67 | 72
T-Score | 46.48 (7.6) | 50.8 (7.4)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | 20 mL 0.5% Bupivacaine HCL | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5%
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/78
Other Adverse Events (participants affected / at risk) | 2/72 | 5/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mL 0.5% Bupivacaine HCL (N=72) | Interscalene Nerve Block With Liposomal + Bupivacaine 0.5% (N=78)
Stress Fracture During Physical Therapy (Musculoskeletal and connective tissue disorders) | 0 | 1
ER visit due to bowel obstruction from opioids (Gastrointestinal disorders) | 1 | 0
Swelling on wrist/fingers 3 weeks post-op (Musculoskeletal and connective tissue disorders) | 0 | 1
Revision surgery required 1 week post-op (Surgical and medical procedures) | 1 | 0
Elevated hemi diaphragm from prolonged phrenic nerve block (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Shoulder dislocation, required additional meds (Musculoskeletal and connective tissue disorders) | 0 | 1
Intra-op fracture (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03913091/Prot_SAP_000.pdf